CLINICAL TRIAL: NCT00318877
Title: Sports to Prevent Obesity Randomized Trial
Brief Title: Sports to Prevent Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31487; 1R03DK070580-01 (NIH)
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Obesity
Keywords: Obesity; Physical activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- After school sports (Experimental): After school team sports
  Interventions: Behavioral: After school team sports program
- Health and Nutrition Education (Active Comparator): Health and Nutrition Education Active Placebo Control
  Interventions: Behavioral: After school health education program

INTERVENTIONS:
Behavioral: After school team sports program
  Arms: After school sports
Behavioral: After school health education program
  Arms: Health and Nutrition Education

SUMMARY:
The purpose of this study is to learn whether overweight children who participate in an after school team sports program improve their health as much as overweight children in a more traditional health education program.

DETAILED DESCRIPTION:
There is an urgent need for feasible, effective, and cost-efficient programs to help overweight children control their weight. To start to address this unmet need, we are evaluating after school team sports as an intervention for reducing weight gain among low-income and at-risk of being overweight, and overweight children. After school sports programs may be generalizable, motivating, and cost-efficient interventions for long-term weight control among at-risk and overweight children. The infrastructure needed to provide such programs already exists in most communities. In contrast, more traditional, medically- and behaviorally-oriented treatment programs are expensive, generally not very effective, often inconvenient, and not available in most communities. While children involved in team sports tend to be more physically fit than their uninvolved peers, team sports has not yet been tested as a method to increase involvement of at-risk and overweight children in regular physical activity. As an added bonus, these sports programs can displace typical after school television viewing and snacking. Team sports is a potentially innovative and high impact approach for intervening with at-risk and overweight children, as it may provide an opportunity to reduce weight gain while increasing social interaction and self-esteem. If our proposed research finds that team sports are an efficacious intervention for reducing weight gain among low-income, at-risk and overweight children, it is an intervention approach that could be rapidly diffused and tested for effectiveness. The policy implications of these findings would be great, encouraging expanded access to team sports programs to a population that has not been previously targeted or included.

We propose a 1 year randomized controlled trial comparing weight changes among low-income, overweight children randomized to participate in an after school team sports program versus a traditional weight control/health education program.

ELIGIBILITY:
Inclusion Criteria:

* In the participating school district
* 8-11.9 years old
* BMI >= 85th percentile for age and sex on the 2000 Centers for Disease Control (CDC) growth charts
* Clearance to participate from medical care provider
* Willing, able, and available to attend an after school program
* Not planning to move from school district within the next 12 months
* Speaks and reads English or Spanish
* Child has not repeated more than one grade in school
* Completion of signed active informed consent (parent or guardian) and assent (child) to participate, which includes a description of the two interventions and requires their willingness to be randomized.

Exclusion Criteria:

The investigators' goal is to be as inclusive as possible, however, children will not be eligible to participate if they:

* Have a condition that limits their participation in physical activity enough that they are not able to participate in Physical Education at school (e.g. significant structural heart disease)
* Have been diagnosed with a chronic illness that affects their growth and/or weight (e.g. type 1 diabetes, hypothyroidism, inflammatory bowel disease)
* Have taken systemic steroids (oral, intravenous, or intramuscular) for a period of more than 21 days in the past year
* Are taking other medications affecting their growth and/or weight [e.g. methylphenidate hydrochloride (HCL)]
* Are pregnant
* Are unable to complete the informed consent process

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2006-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | baseline to follow-up

SECONDARY OUTCOMES:
Waist circumference | baseline to follow-up
Triceps skinfold thickness | baseline to follow-up
Resting heart rate | baseline to follow-up
Blood pressure | baseline to follow-up
Physical activity monitoring | baseline to follow-up
Sedentary behaviors | baseline to follow-up
Psychosocial measures | baseline to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Robinson, MD, MPH, Principal Investigator — Stanford University; Dana L Weintraub, MD, Study Director — Stanford University
Locations (1):
- Stanford Prevention Research Center, Palo Alto, California, United States